CLINICAL TRIAL: NCT07076368
Title: Determination of the 90% Effective Volume (ED90) of Epidural 0.1% Ropivacaine and Fentanyl for Labor Analgesia Initiation in Patients Receiving a Dural-Puncture Epidural Technique
Brief Title: Ropivacaine and Fentanyl for Labor Epidural Initiation
Acronym: EV90_DPE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-43988
Record Dates: First submitted 2025-07-07; First posted 2025-07-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Labor and Delivery; Labor Analgesia
Keywords: epidural; labor analgesia; pregnancy; obstetric anesthesia
MeSH Terms: interventions — Ropivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: This is a single-center, double-blind, prospective study that will use a biased-coin-up-down allocation study design to quantify the effective volume in 90% of laboring patients (EDV) after a dural-puncture epidural (DPE) technique for neuraxial analgesia. We wish to declare that the participant, care providers, and outcomes assessor will be masked. The ClinicalTrials website does not allow us to tick these roles for a single-arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Observational Cohort (Experimental): Patients with singleton vertex pregnancies in active labor (spontaneous or after induction of labor), with a cervical dilatation between 1 and 7cm who are requesting neuraxial labor analgesia, Age =>18 yrs
  Interventions: Drug: Ropivacaine + Fentanyl

INTERVENTIONS:
Drug: Ropivacaine + Fentanyl — A standard epidural admixture - 0.1% Ropivacaine + 2 mcg/ml fentanyl - will be used.

SUMMARY:
This study is being done to determine the most effective dose of medicine to use to initially provide effective pain relief within the first 30 minutes of receiving an epidural for pain labor during labor. The study team will also study any side effects related to the epidural medication and patients' satisfaction with the quality of pain relief after receiving the epidural.

DETAILED DESCRIPTION:
We aim to perform a prospective observational study in a single cohort of 50 patients receiving a dural-puncture epidural technique for labor analgesia. We will use a biased-coin up-down allocation methodology to quantify the volume of a combined epidural 0.1% ropivacaine and 2 mcg/ml fentanyl regimen that achieves effective analgesia in 90% of patients experiencing active labor who receive a dural-puncture epidural technique for labor analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with singleton vertex pregnancies in active labor (latent or spontaneous labor or after induction of labor)
* Cervical dilatation between 2 and 7 cm
* Requesting neuraxial labor analgesia
* Age 18 or older

Exclusion Criteria:

* Significant obstetric disease (e.g., pre-eclampsia, major cardiac disease)
* Chronic pain or chronic opioid use
* BMI ≥ 50
* Multiple gestations
* Allergy or anaphylaxis to local anesthetic
* Fetal compromise or non-reassuring fetal trace
* Age under 18
* Inability to speak and understand English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant birthing patients
Enrollment: 50 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain score | 30 mins post-intervention
  Numerical pain score using a discrete range from 0 (no pain) to 10 (most severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Butwick, MBBS, FRCA, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707
- [Background] Song Y, Song Y, Sheng Z, Zhao Q, Liu W, Li Y, Zang Y, Xu Z, Liu Z. Exploration of the optimal programmed intermittent epidural bolus volume with the dural puncture epidural technique for labour analgesia: a biased-coin up-and-down sequential allocation study. Can J Anaesth. 2025 Feb;72(2):254-261. doi: 10.1007/s12630-024-02855-6. Epub 2024 Oct 21. PMID 39433721
- [Background] Maeda A, Villela-Franyutti D, Lumbreras-Marquez MI, Murthy A, Fields KG, Justice S, Tsen LC. Labor Analgesia Initiation With Dural Puncture Epidural Versus Conventional Epidural Techniques: A Randomized Biased-Coin Sequential Allocation Trial to Determine the Effective Dose for 90% of Patients of Bupivacaine. Anesth Analg. 2024 Jun 1;138(6):1205-1214. doi: 10.1213/ANE.0000000000006691. Epub 2023 Oct 12. PMID 37824436